CLINICAL TRIAL: NCT02280408
Title: A Phase 1 Randomized, Double-Blind, Placebo Controlled, Dose-Escalation Study to Evaluate the Safety and Immunogenicity of Prime-Boost VSV Ebola Vaccine in Healthy Adults
Brief Title: Safety and Immunogenicity of Prime-Boost Vesicular Stomatitis Virus (VSV) Ebola Vaccine in Healthy Adults (V920-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); BioProtection Systems Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V920-002; NLG0207 (Study 15-I-0001) (Other: NewLink Genetics Corp.)
Record Dates: First submitted 2014-10-23; First posted 2014-10-31 (Estimated); Results first posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Ebola Viruses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 3x10^6 plaque-forming units (pfu) Vaccine Cohort (Experimental): Participants will receive a 1-mL intramuscular injection of V920 3x10^6 pfu in the deltoid on Day 0 and Day 28.
  Interventions: Biological: V920
- 2x10^7 pfu Vaccine Cohort (Experimental): Participants will receive a 1-mL intramuscular injection of V920 2x10^7 pfu in the deltoid on Day 0 and Day 28.
  Interventions: Biological: V920
- 1x10^8 pfu Vaccine Cohort (Experimental): Participants will receive a 1-mL intramuscular injection of V920 1x10^8 pfu in the deltoid on Day 0 and Day 28.
  Interventions: Biological: V920
- Placebo Cohort (Placebo Comparator): Participants will receive a 1-mL intramuscular injection of placebo in the deltoid on Day 0 and Day 28.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Normal saline placebo.
  Arms: Placebo Cohort
Biological: V920 — Vesicular Stomatitis Virus (VSV)-based vaccine 1-mL injection containing 3x10^6, 2x10^7, or 1x10^8 pfu.
  Arms: 1x10^8 pfu Vaccine Cohort; 2x10^7 pfu Vaccine Cohort; 3x10^6 plaque-forming units (pfu) Vaccine Cohort

SUMMARY:
Ebola virus has infected and killed people, mostly in Africa. In 2014, the Zaire ebolavirus (ZEBOV) has affected several thousand people. There is no approved effective way to treat or prevent Ebola. Researchers are trying to develop a vaccine for it. This is a study of the anti-Ebola vaccine vesicular stomatitis virus (VSV) ZEBOV (V920; BPSC-1001) to see if it is safe and to see how it affects people's immune system.

DETAILED DESCRIPTION:
Between 1994 and the present, there have been many Ebola virus (EBOV) outbreaks affecting mostly central Africa. However, the 2014 West African outbreak significantly exceeds all previous outbreaks in geographic range, number of individuals affected and in disruption of typical activities of civil society.

This is a Phase 1 safety and tolerability study to evaluate a novel vaccine to Ebola using a live VSV replacing the gene encoding the G envelope glycoprotein with the gene encoding the envelope glycoprotein from the Zaire strain of Ebola (VSVΔG-ZEBOV also known as V920 and BPSC-1001).

ELIGIBILITY:
INCLUSION CRITERIA:

* Healthy male or females, ages 18 to 65 (inclusive) at the time of screening
* Females of childbearing potential and all males, must be willing to use effective methods of contraception, from at least 14 days prior to vaccination through Day 56 which would include:

  * Oral contraceptives, either combined or progestogen alone
  * injectable progestogen
  * implants of etonogestrel or levonorgestrel
  * oestrogenic vaginal ring
  * percutaneous contraceptive patches
  * intrauterine device or intrauterine system
  * male partner sterilization
  * male condom combined with a spermicide
* Must be willing to minimize blood and body fluid exposure of others for at least 7 days after vaccination, which includes:

  * Use of effective barrier prophylaxis, such as latex condoms, during any sexual interaction (regardless of childbearing status or sexual orientation)
  * Avoiding the sharing of needles, razors, eating utensils, drinking from the same cup, or toothbrushes
  * Avoiding open-mouth kissing
* Must be willing to forgo blood donation for one year
* Must agree not to enroll in another study of an investigational agent prior to completion of Day 56 and not participate in an investigational vaccine study until the last required protocol visit on Day 365
* Ability to provide informed consent

EXCLUSION CRITERIA:

FACTORS THAT INCREASE RISK TO THE SUBJECT:

* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response
  * A process that would require medication that affects the immune response
  * Any contraindication to repeated injections or blood draws
  * A condition that requires active medical intervention or monitoring to avert grave danger to the participant's health or well-being during the study period
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine
  * Any condition specifically listed among the exclusion criteria below
  * Active malignancy
  * Asplenia
  * History of Guillain-Barré Syndrome
  * History of neurological or neuropsychiatric disorder that may either increase risk (history of encephalitis, narcolepsy, stroke, depression, bipolar disorder, seizure, etc.) or could interfere with the assessment of safety (e.g., frequent headaches)
  * History of autoimmune disease
  * History of hemoglobinopathy or a coagulopathy
* Women who are breast-feeding
* Positive urine or serum pregnancy test
* Abnormal chemistry panel; defined as:

  * Defined as any Grade 3 or greater toxicity (regardless of clinical significance) by the toxicity table
  * Evaluating only creatinine, alanine aminotransferase, aspartate aminotransferase, total bilirubin, and estimated glomerular filtration rate
* Abnormal complete blood count (CBC) defined as:

  * Defined as any Grade 3 or greater toxicity (regardless of clinical significance) by the toxicity table
  * Evaluating only the white blood cell (WBC), hemoglobin, hematocrit, and platelets
* Abnormal urinalysis defined as:

  * Defined as any Grade 3 or greater toxicity (regardless of clinical significance) by the toxicity table
  * Evaluating red blood cells (RBC), protein, and glucose only
* Positive serology for hepatitis B surface antigen
* Positive serology for hepatitis C
* Positive serology for human immunodeficiency virus (HIV)
* Known allergy to the components of the VSVΔG-ZEBOV vaccine (V920) vaccine product (VSV, albumin, tris)
* History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions

FACTORS THAT MAY LIMIT VSV REPLICATION OR MAKE INTERPRETATION OF IMMUNOGENICITY DIFFICULT:

* History of prior infection with a filovirus or prior participation in a filovirus vaccine trial
* Veterinarian or ranchers exposed to livestock known to be infected with VSV
* History of prior infection with VSV or receipt of a VSV vectored vaccine

FACTORS THAT WOULD INCREASE RISK TO OTHERS DUE TO VSV VIRAL SHEDDING:

* Is a healthcare worker who will have direct contact with patients within 14 days of each vaccination
* Is an animal care worker, who will have direct contact with animals (livestock or domestic, besides subjects family pet) within 14 days of each vaccination
* Has a house-hold contact (HHC) who is immunodeficient (in the opinion of the investigator), pregnant, has an unstable medical condition, or is under the age of 5 years
* Is a childcare worker who has direct contact with children 5 years of age or younger

FACTORS THAT COULD IMPAIR INTERPRETATION OR EXECUTION OF THE STUDY:

* Receipt of any investigational drug within 5 half-lives or 30 days, whichever is longer, prior to study drug administration (i.e., Day 0)
* Receipt of licensed vaccines 14 days before the planned study immunization
* Receipt of immunoglobulins and/or any blood products within the 120 days preceding study entry or that are planned during the study period
* Immunosuppressive medications received within 168 days before first vaccination. (Not including: [1] corticosteroid nasal spray for allergic rhinitis; [2] topical corticosteroids for mild, uncomplicated dermatitis; or [3] oral/parenteral corticosteroids given for non-chronic conditions not expected to recur [length of therapy 10 days or less with completion at least 30 days prior to vaccination(s)].)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled through Day 56
* Participants who, in the judgment of the investigator, will be unlikely to comply with the requirements of this protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-10-07 (Actual); Primary Completion 2015-12-10 (Actual); Study Completion 2015-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Coller BG, Blue J, Das R, Dubey S, Finelli L, Gupta S, Helmond F, Grant-Klein RJ, Liu K, Simon J, Troth S, VanRheenen S, Waterbury J, Wivel A, Wolf J, Heppner DG, Kemp T, Nichols R, Monath TP. Clinical development of a recombinant Ebola vaccine in the midst of an unprecedented epidemic. Vaccine. 2017 Aug 16;35(35 Pt A):4465-4469. doi: 10.1016/j.vaccine.2017.05.097. Epub 2017 Jun 21. PMID 28647166
- [Derived] Regules JA, Beigel JH, Paolino KM, Voell J, Castellano AR, Hu Z, Munoz P, Moon JE, Ruck RC, Bennett JW, Twomey PS, Gutierrez RL, Remich SA, Hack HR, Wisniewski ML, Josleyn MD, Kwilas SA, Van Deusen N, Mbaya OT, Zhou Y, Stanley DA, Jing W, Smith KS, Shi M, Ledgerwood JE, Graham BS, Sullivan NJ, Jagodzinski LL, Peel SA, Alimonti JB, Hooper JW, Silvera PM, Martin BK, Monath TP, Ramsey WJ, Link CJ, Lane HC, Michael NL, Davey RT Jr, Thomas SJ; rVSVDeltaG-ZEBOV-GP Study Group. A Recombinant Vesicular Stomatitis Virus Ebola Vaccine. N Engl J Med. 2017 Jan 26;376(4):330-341. doi: 10.1056/NEJMoa1414216. Epub 2015 Apr 1. PMID 25830322

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Started | 10 | 10 | 10 | 9
Vaccination 1 | 10 | 10 | 10 | 9
Vaccination 2 | 10 | 10 | 10 | 9
Completed | 10 | 8 | 10 | 9
Not Completed | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort | Total
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 9 | 39
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 3 | 3 | 11
  Male | 6 | 9 | 7 | 6 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 1 or More Unsolicited AE : Vaccination 1
Description: An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study drug or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study vaccine or protocol-specified procedure is also an AE. An unsolicited AE was an AE other than those specifically designated local or systemic. The percentage of participants that experienced at least 1 unsolicited AE was summarized.
Time Frame: Up to 28 days post vaccination 1 (From Day 1 up to Day 28)
Population: All randomized participants who received at least 1 vaccination with V920 or placebo and had follow-up data for endpoint
Measure: Number; unit: Percentage of participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Percentage of participants | 60.0 | 70.0 | 50.0 | 44.4

2. Primary Outcome: Percentage of Participants With 1 or More Unsolicited AE : Vaccination 2
Description: as for outcome 1
Time Frame: Up to 28 days post vaccination 2 (From Day 29 to Day 56)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Percentage of participants | 70.0 | 50.0 | 90.0 | 44.4

3. Primary Outcome: Percentage of Participants With 1 or More Solicited Systemic Adverse Event (AE) by Severity: Vaccination 1
Description: A solicited AE was a predetermined specific event. The solicited systemic AEs for this study were the following: redness, swelling, or pain at site of injection, subjective and objective fever, chills, sweats, myalgia, arthralgia, fatigue, headache and gastrointestinal symptoms (nausea, vomiting, abdominal pain, and/or diarrhea). All AEs were assessed for severity by the investigator according to the Food and Drug Administration(FDA's) Guidance "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" and were classified into 4 categories: Mild (Grade 1), Moderate (Grade 2), Severe (Grade 3) and Potentially Life-Threatening (Grade 4). The percentage of participants that experienced at least 1 solicited systemic AE were summarized by grade.
Time Frame: Up to 14 days post vaccination 1 (From Day 1 up to Day 14)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Percentage of Participants
  Mild (Grade 1) | 40.0 | 40.0 | 10.0 | 22.2
  Moderate (Grade 2) | 50.0 | 60.0 | 60.0 | 11.1
  Severe (Grade 3) | 10.0 | 0.0 | 10.0 | 0.0
  Life-threatening (Grade 4) | 0.0 | 0.0 | 0.0 | 0.0

4. Primary Outcome: Percentage of Participants With 1 or More Solicited Systemic AE by Severity: Vaccination 2
Description: as for outcome 3
Time Frame: Up to 14 days post vaccination 2 (Day 29 up to Day 42)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Percentage of Participants
  Mild (Grade 1) | 30.0 | 40.0 | 20.0 | 0.0
  Moderate (Grade 2) | 10.0 | 10.0 | 20.0 | 11.1
  Severe (Grade 3) | 0.0 | 0.0 | 10.0 | 0.0
  Life-threatening (Grade 4) | 0.0 | 0.0 | 0.0 | 0.0

5. Primary Outcome: Percentage of Participants With One or More Serious Adverse Event
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the study vaccine. An SAE is an AE that results in death, is life-threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, or is another important medical event. The percentage of participants that experienced 1 or more SAEs was summarized.
Time Frame: Up to Day 56 (Day 1 up to Day 56)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

6. Primary Outcome: Percentage of Participants With 1 or More Solicited Local Injection-site AE by Severity: Vaccination 1
Description: A solicited AE was a predetermined specific event. The solicited local AEs for this study were the following: Local reactogenicity signs and symptoms include pain, erythema (redness), and induration (swelling). All AEs were assessed for severity by the investigator according to the Food and Drug Administration(FDA's) Guidance "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" and were classified into 4 categories: Mild (Grade 1), Moderate (Grade 2), Severe (Grade 3) and Potentially Life-Threatening (Grade 4). The percentage of participants that experienced at least 1 solicited local AE was summarized by grade.
Time Frame: Up to 14 days post vaccination 1 (Day 1 to Day 14)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Percentage of participants
  Mild (Grade 1) | 60.0 | 80.0 | 60.0 | 11.1
  Moderate (Grade 2) | 10.0 | 20.0 | 20.0 | 0.0
  Severe (Grade 3) | 0.0 | 0.0 | 0.0 | 0.0
  Life-threatening (Grade 4) | 0.0 | 0.0 | 0.0 | 0.0

7. Primary Outcome: Percentage of Participants With 1 or More Solicited Local Injection-site AE by Severity: Vaccination 2
Description: as for outcome 6
Time Frame: Up to 14 days post vaccination 2 (Day 29 up to Day 42)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Percentage of participants
  Mild (Grade 1) | 30.0 | 80.0 | 70.0 | 44.4
  Moderate (Grade 2) | 0.0 | 0.0 | 10.0 | 0.0
  Severe (Grade 3) | 0.0 | 0.0 | 0.0 | 0.0
  Life-threatening (Grade 4) | 0.0 | 0.0 | 0.0 | 0.0

8. Primary Outcome: Percentage of Participants With Early Discontinuation of Vaccination
Description: The percentage of participants that had vaccination discontinued for any reason was summarized.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

9. Secondary Outcome: Geometric Mean Titers of Zaire Ebolavirus-(ZEBOV)-Specific Immunoglobin G (IgG) Antibodies: Day 28
Description: Blood was drawn on Day 28 to assess the GMTs of ZEBOV-specific IgG antibodies as determined by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 28
Population: All randomized participants who were vaccinated twice with V920 or placebo, had ZEBOV IgG ELISA endpoint titer results on Days 0 (baseline) and 28, and who did not have any protocol violations that influenced interpretation of immunogenicity endpoints.
Measure: Geometric Mean (Standard Deviation); unit: ELISA Units/mL
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
ELISA Units/mL | 897.61 (3.26) | 2506.03 (2.67) | 2469.07 (1.82) | 29.42 (1.00)
Statistical Analysis 1: Comparison: 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort vs Placebo Cohort; Test type: Other; p < 0.001, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 2: Comparison: 2x10^7 Pfu Vaccine Cohort vs Placebo Cohort; Test type: Other; p < 0.001, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 3: Comparison: 1x10^8 Pfu Vaccine Cohort vs Placebo Cohort; Test type: Other; p < 0.001, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 4: Comparison: 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort vs 2x10^7 Pfu Vaccine Cohort; Test type: Other; p = 0.010, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 5: Comparison: 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort vs 1x10^8 Pfu Vaccine Cohort; Test type: Other; p = 0.011, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 6: Comparison: 2x10^7 Pfu Vaccine Cohort vs 1x10^8 Pfu Vaccine Cohort; Test type: Other; p = 0.969, ANOVA; Adjustments for multiple comparisons were not performed

10. Secondary Outcome: Geometric Mean Titers of ZEBOV-specific IgG Antibodies: Day 56
Description: Blood was drawn on Day 56 to assess the GMTs of ZEBOV-specific IgG antibodies as determined by Enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 56 (28 days post vaccination 2)
Population: All randomized participants who were vaccinated twice with V920 or placebo, had ZEBOV IgG ELISA endpoint titer results on Days 0 (baseline) and 56, and who did not have any protocol violations that influenced interpretation of immunogenicity endpoints.
Measure: Geometric Mean (Standard Deviation); unit: ELISA Units/mL
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
ELISA Units/mL | 2149.43 (2.07) | 5320.73 (1.50) | 5710.33 (1.42) | 29.42 (1.00)
Statistical Analysis 1: Comparison: 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort vs Placebo Cohort; Test type: Other; p < 0.001, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 2: Comparison: 2x10^7 Pfu Vaccine Cohort vs Placebo Cohort; Test type: Other; p < 0.001, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 3: Comparison: 1x10^8 Pfu Vaccine Cohort vs Placebo Cohort; Test type: Other; p < 0.001, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 4: Comparison: 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort vs 2x10^7 Pfu Vaccine Cohort; Test type: Other; p < 0.001, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 5: Comparison: 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort vs 1x10^8 Pfu Vaccine Cohort; Test type: Other; p < 0.001, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 6: Comparison: 2x10^7 Pfu Vaccine Cohort vs 1x10^8 Pfu Vaccine Cohort; Test type: Other; p = 0.733, ANOVA; Adjustments for multiple comparisons were not performed

11. Secondary Outcome: Geometric Mean Titers of ZEBOV-specific Neutralizing Antibodies: Day 28
Description: Blood was drawn on Day 28 to assess the GMTs of Zaire ebolavirus neutralizing antibodies as determined by Pseudovirion neutralizing assay (PsVNA). Titers are reported for PsVNA50 values, which was derived from the reciprocal of the dilution that resulted in a 50% decrease in luciferase activity.
Time Frame: Day 28 (28 days post vaccination 1)
Population: as for outcome 9
Measure: Geometric Mean (Standard Deviation); unit: Titer
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Titer | 222.2 (1.91) | 415.8 (3.93) | 475.5 (2.61) | 10.0 (1.00)
Statistical Analysis 1: Comparison: 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort vs Placebo Cohort; Test type: Other; p < 0.001, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 2: Comparison: 2x10^7 Pfu Vaccine Cohort vs Placebo Cohort; Test type: Other; p < 0.001, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 3: Comparison: 1x10^8 Pfu Vaccine Cohort vs Placebo Cohort; Test type: Other; p < 0.001, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 4: Comparison: 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort vs 2x10^7 Pfu Vaccine Cohort; Test type: Other; p = 0.132, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 5: Comparison: 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort vs 1x10^8 Pfu Vaccine Cohort; Test type: Other; p = 0.070, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 6: Comparison: 2x10^7 Pfu Vaccine Cohort vs 1x10^8 Pfu Vaccine Cohort; Test type: Other; p = 0.743, ANOVA; Adjustments for multiple comparisons were not performed

12. Secondary Outcome: Geometric Mean Titers of ZEBOV-specific Neutralizing Antibodies: Day 56
Description: Blood was drawn on Day 56 to assess the GMTs of Zaire ebolavirus neutralizing antibodies as determined by Pseudovirion neutralizing assay (PsVNA). Titers are reported for PsVNA50 values, which was derived from the reciprocal of the dilution that resulted in a 50% decrease in luciferase activity.
Time Frame: Day 56 (28 days post vaccination 2)
Population: as for outcome 10
Measure: Geometric Mean (Standard Deviation); unit: Titer
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Titer | 344.1 (2.09) | 653.0 (1.59) | 669.0 (1.93) | 10.0 (1.00)
Statistical Analysis 1: Comparison: 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort vs Placebo Cohort; Test type: Other; p < 0.001, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 2: Comparison: 2x10^7 Pfu Vaccine Cohort vs Placebo Cohort; Test type: Other; p < 0.001, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 3: Comparison: 1x10^8 Pfu Vaccine Cohort vs Placebo Cohort; Test type: Other; p < 0.001, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 4: Comparison: 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort vs 2x10^7 Pfu Vaccine Cohort; Test type: Other; p = 0.014, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 5: Comparison: 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort vs 1x10^8 Pfu Vaccine Cohort; Test type: Other; p = 0.011, ANOVA; Adjustments for multiple comparisons were not performed
Statistical Analysis 6: Comparison: 2x10^7 Pfu Vaccine Cohort vs 1x10^8 Pfu Vaccine Cohort; Test type: Other; p = 0.923, ANOVA; Adjustments for multiple comparisons were not performed

13. Secondary Outcome: Percentage of Participants Who Seroconvert: Day 28
Description: GMTs for Zebov-specific antibodies were determined via ELISA. Seroconversion was defined as a post-vaccination titer ≥ 200 that is also at least a 4-fold increase in titer compared to baseline.
Time Frame: Day 28 (28 days post vaccination 1)
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Percentage of Participants | 100.0 | 100.0 | 100.0 | 0.0

14. Secondary Outcome: Percentage of Participants Who Seroconvert: Day 56
Description: as for outcome 13
Time Frame: Day 56 (28 days post vaccination 2)
Population: as for outcome 10
Measure: Number; unit: Percentage of Participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Percentage of Participants | 100.0 | 100.0 | 100.0 | 0.0

15. Secondary Outcome: Percentage of Participants With Viremia on Day 3 and Day 7: Vaccination 1
Description: Blood was drawn on Days 3 and 7 to assess the presence of V920 via polymerase chain reaction (PCR) assay. The percentage of participants that were positive for V920 in serum was summarized.
Time Frame: Day 3 and Day 7 post vaccination 1
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Percentage of Participants
  Day 3 post vaccination 1 | 100.0 | 100.0 | 100.0 | 0.0
  Day 7 post vaccination 1 | 0.0 | 30.0 | 30.0 | 0.0

16. Secondary Outcome: Percentage of Participants With Viremia on Day 3 and Day 7: Vaccination 2
Description: as for outcome 15
Time Frame: Day 3 and Day 7 post vaccination 2 (Day 31 and Day 35)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Percentage of Participants
  Day 3 post vaccination 2 | 0.0 | 0.0 | 12.5 | 0.0
  Day 7 post vaccination 2 | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: up to Day 365 (approximately 1 years post vaccination 1)
Description: All participants that received at least 1 study vaccination and had follow-up safety data.
Groups:
- 3x106 Pfu V920: Participants will receive a 1-mL intramuscular injection of V920 3x10^6 pfu in the deltoid on Day 0 and Day 28.
- 2x107 Pfu V920: Participants will receive a 1-mL intramuscular injection of V920 2x10^7 pfu in the deltoid on Day 0 and Day 28.
- 1x108 Pfu V920: Participants will receive a 1-mL intramuscular injection of V920 1x10^8 pfu in the deltoid on Day 0 and Day 28.
- Placebo: Participants will receive a 1-mL intramuscular injection of placebo in the deltoid on Day 0 and Day 28.
Arm/Group | 3x106 Pfu V920 | 2x107 Pfu V920 | 1x108 Pfu V920 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 10/10 | 8/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3x106 Pfu V920 (N=10) | 2x107 Pfu V920 (N=10) | 1x108 Pfu V920 (N=10) | Placebo (N=9)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (6) | 2 (2) | 1 (2)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 5 (6) | 7 (8) | 5 (5) | 0 (0)
Fatigue (General disorders) | 7 (11) | 9 (13) | 7 (12) | 2 (4)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 7 (12) | 8 (17) | 4 (11) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 2 (5) | 2 (3) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1) | 2 (3) | 1 (1)
Lymphocyte percentage decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (3) | 2 (3) | 4 (5) | 2 (2)
Prothrombin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 2 (3) | 1 (2) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (9) | 6 (11) | 4 (6) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (11) | 10 (14) | 6 (12) | 2 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 8 (15) | 7 (10) | 5 (10) | 1 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glycosuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (7) | 2 (3)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No